CLINICAL TRIAL: NCT04340466
Title: French Multicentre Observational Study on SARS-Cov-2 Infections (COVID-19) ICU Management: the FRENCH CORONA Study
Brief Title: French Multicentre Observational Study on SARS-Cov-2 Infections (COVID-19) ICU Management Study
Acronym: FRENCH CORONA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00797-32; 2020-A00797-32 (Other: ANSM)
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2020-12

CONDITIONS: Pneumonia, Viral; Critically Ill; Corona Virus Infection
Keywords: COVID-19; SARS-Cov-2; Intensive Care Unit
MeSH Terms: conditions — Pneumonia, Viral; Critical Illness; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected or proven COVID-19 critically ill patients
  Interventions: Other: No intervention
- Control
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Since December 2019, a new agent, the SARS-Cov-2 coronavirus has been rapidly spreading from China to other countries causing an international outbreak of respiratory illnesses named COVID-19. In France, the first cases have been reported at the end of January with more than 60000 cases reported since then. A significant proportion (20-30%) of hospitalized COVID-19 patients will be admitted to intensive care unit. However, few data are available for this special population in France.

We conduct a large observational cohort of ICU suspected or proven COVID-19 patients that will enable to describe the initial management of COVID 19 patients admitted to ICU and to identify factors correlated to clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU for suspected or proven SARS-Cov-2 infection, defined by positive SARS-Cov-2 PCR or CT scan images
* Patient > or= 18 years

Exclusion Criteria:

* Patient study refusal
* Patient already enrolled in the present study
* Patient with respiratory illness with negative COVID-19 CT scan images and negative COVID_19 PCR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study is all patients with suspected or proven SARS-Cov-2 infection (COVID-19)
Sampling Method: Non-Probability Sample
Enrollment: 1003 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Mortality at day 28 | day 28
  Mortality at day 28

SECONDARY OUTCOMES:
severe complications | up to day 28
  severe complications (pulmonary embolism, acute kidney injury, myocarditis, cardiac arrest, liver failure, ventilator associated pneumonia) Yes / No
Imaging | day 1
  Delay in imaging in hours
Delay in Microbiological diagnosis | day 1
  delay in microbiological diagnosis in hours
Antiviral therapy | up to day 28
  Antiviral therapy Yes / no
Antibiotic therapy | day 28
  Antibiotic therapy Yes / No
Covid-19 treatments | up to day 28
  Covid-19 treatments Yes / No
Patients receiving renal replacement therapy | up to day 28
  number
Patients receiving mechanical ventilation | up to day 28
  number
Vital status | day 28
  Patient alive at day 28 : yes / No

CONTACTS AND LOCATIONS:
Overall Officials: CLAIRE ROGER, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Roger C, Collange O, Mezzarobba M, Abou-Arab O, Teule L, Garnier M, Hoffmann C, Muller L, Lefrant JY, Guinot PG, Novy E, Abraham P, Clavier T, Bourenne J, Besch G, Favier L, Fiani M, Ouattara A, Joannes-Boyau O, Fischer MO, Leone M, Ait Tamlihat Y, Pottecher J, Cordier PY, Aussant P, Moussa MD, Hautin E, Bouex M, Julia JM, Cady J, Danguy Des Deserts M, Mayeur N, Mura T, Allaouchiche B; AZUREA group. French multicentre observational study on SARS-CoV-2 infections intensive care initial management: the FRENCH CORONA study. Anaesth Crit Care Pain Med. 2021 Aug;40(4):100931. doi: 10.1016/j.accpm.2021.100931. Epub 2021 Jul 10. PMID 34256165